CLINICAL TRIAL: NCT05174650
Title: A Phase II Single-arm, Open-label Study of Atezolizumab and Derazantinib for Patients With Advanced Intrahepatic Cholangiocarcinoma With FGFR2
Brief Title: Treatment of Atezolizumab and Derazantinib in Patients With Advanced iCCA With FGFR2 Fusions/Rearrangements
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institut für Klinische Krebsforschung IKF GmbH at Krankenhaus Nordwest (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ADVANCE_2020
Record Dates: First submitted 2021-11-09; First posted 2022-01-03 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-04

CONDITIONS: Intrahepatic Cholangiocarcinoma
MeSH Terms: conditions — Cholangiocarcinoma | interventions — atezolizumab; derazantinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Combined treatment with Atezolizumab and Derazantinib (Experimental): Treatment with Atezolizumab 1200 mg i.v. every 3 weeks and Derazantinib 300 mp p.o. once daily for a maximum of 60 weeks or until disease progression or unacceptable toxicity or study termination
  Interventions: Drug: Atezolizumab; Drug: Derazantinib

INTERVENTIONS:
Drug: Atezolizumab — Infusion i.v. of atezolizumab on day 1 of a 3-week cycle, first infusion rate over 60 minutes, subsequent infusion rates 30 minutes if tolerated for a maximum of 20 cycles in total
  Other Names: Tecentriq
Drug: Derazantinib — Oral intake of 300 mg derazantinib continuously on day 1 to day 21 of a 3-week cycle for a maximum of 20 cycles in total
  Other Names: ARQ 087

SUMMARY:
The study trial is a open-label, single-arm, multicenter phase II trial investigating the combined treatment of atezolizumab and derazantinib in patients with advanced intrahepatic cholangiocarcinoma with FGFR2 fusions/rearrangements

DETAILED DESCRIPTION:
The aim of this phase II study is to explore the safety and anti-tumor efficacy of the combination of atezolizumab and derazantinib in patients with advanced intrahepatic cholangiocarcinoma, with ORR as the primary endpoint.

The primary endpoint is the Objective Response Rate (ORR [assessed every 8 weeks (±7 days)]):

Objective response rate (ORR) according to investigator-based RECIST 1.1 assessment, defined as the proportion of allocated subjects with best response of complete or partial response within 9 months after the date of first administration of study treatment.

The secondary endpoints are safety and efficacy and will be evaluated by

* Incidence, treatment relationship, seriousness, and severity of all AEs, SAEs, AESIs according to CTCAE V5.0
* ORR@EOT:

Objective response rate (ORR) according to investigator-based RECIST 1.1 assessment, defined as the proportion of allocated subjects with best response of complete or partial response within study treatment.

• PFSR@6, 8 and 10 months: The proportion of patients known to be alive and without confirmed objective disease progression at 6, 8 and 10 months after first administration of study treatment, respectively.

• PFS: Time from first administration of study treatment until the date of first objective disease progression or death.

• OS: Time from first administration of study treatment until death of a patient due to any cause

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all of the following criteria to be eligible for the study:

1. Fully informed written consent and locally required authorization (European Union [EU] Data Privacy Directive in the EU) obtained from the patient prior to performing any protocol-related procedures, including screening evaluations.
2. Patients*, age ≥ 18 years at the time of signing the Informed Consent Form.
3. Histologically documented diagnosis of non-resectable iCCA with positively confirmed FGFR2 fusion/rearrangement via NGS-Analysis.

   Note: Only CE-IVD marked NGS-tests are applicable which cover FGFR2 fusions and rearrangements.
4. Performance status (PS) ≤ 2 (ECOG scale).
5. At maximum one previous line of systemic anti-cancer therapy, (chemotherapy, hormonal, targeted therapy, experimental therapy) for which treatment was discontinued at least 4 weeks before the first dose of study treatment, or five half-lives of the respective anti-cancer therapy, whichever is the longer period.

   Note: For mABs in previous therapy the restriction to five half-lives does not apply.
6. No prior treatment with any FGFR or immune checkpoint inhibitor (including but not limited to antiCTLA-4, antiPD-1, and antiPD-L1 therapeutic antibodies) apart from Durvalumab as PD-L1 inhibitor in first line therapy.
7. Body weight > 30 kg AND BMI ≥ 15.
8. At least one measurable site of disease as defined by RECIST 1.1 criteria.
9. Adequate bone marrow and renal function including the following:

   * Hemoglobin ≥ 9.0 g/dL (previous transfusion permitted);
   * Absolute neutrophil count (ANC) ≥ 1.500 per µL (1.5×109/L);
   * Platelet count ≥ 75,000 per µL (75 × 109/L);
   * International normalized ratio (INR) between 0.8 × ULN to 1.0 × ULN OR ≤ 3 × ULN for subjects receving anticoagulant therapy
   * Creatinine ≤ 1.5 × ULN OR CLCR ≥ 50 mL/min (as calculated by the Cockcroft-Gault formula);
   * serum phosphate ≤ ULN;
   * corrected serum calcium ≥ 1.75 mmol/L (≥ 7.0 mg/dL) AND ≤ 3.1 mmol/L (≤ 12.5 mg/dL);
   * serum sodium ≥ LLN.
10. Adequate hepatic function (with stenting for any obstruction, if required) including the following:

    o Total bilirubin ≤ 2 × ULN;
    * AST or ALT ≤ 3 × ULN (or ≤ 5 × ULN for subjects with liver metastases);
    * Prothrombin time ≥ 60%;
    * Albumin ≥ 2.8 g/dL.
11. For patients with active hepatitis B virus (HBV):

    * HBV DNA ≤ 500 IU/mL obtained within 28 days prior to initiation of study treatment, AND
    * Anti-HBV treatment (per local standard of care; e.g., entecavir) prior to study entry and willingness to continue treatment for the length of the study.
12. For patients with active hepatitis C virus (HCV):

    * Patients positive for hepatitis C virus (HCV) antibody are eligible, also if polymerase chain reaction testing is positive for HCV ribonucleic acid (RNA).
    * However, anti-viral therapy against HCV is only allowed prior to trial but not during the trial.
13. Negative HIV test.
14. Negative pregnancy test within 72 h prior to dosing.
15. Females of childbearing potential must agree to remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods that result in a failure rate of < 1% per year during the treatment period and for at least 5 months or for a period of at least 5 half-lives of the respective drug/IMP (whichever is longer) after the last study treatment. A woman is considered to be of childbearing potential if she is postmenarcheal, has not reached a postmenopausal state (has not had ≥ 12 continuous months of amenorrhea with no identified cause other than menopause), and has not undergone surgical sterilization (removal of ovaries and/or uterus). Examples of contraceptive methods with a failure rate of < 1% per year include bilateral tubal ligation, male sterilization, hormonal implants, established, proper use of combined oral or injected hormonal contraceptives, and certain intrauterine devices. The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not acceptable methods of contraception.
16. With female partners of childbearing potential, men must remain abstinent or use a condom plus an additional contraceptive method that together result in a failure rate of 1% per year from screening to 5 months after the last dose of combination therapy or for a period of at least 5 half-lives of the respective drug/IMP after the last dose of combination therapy (whichever is longer). Men must refrain from donating sperm during this same period. Men with a pregnant partner must agree to remain abstinent or to use a condom for the duration of the pregnancy to avoid exposing the embryo.
17. The patient is willing and able to comply with the protocol for the duration of the study, including hospital visits for treatment and scheduled follow-up visits and examinations.
18. Must have a life expectancy of at least 12 weeks. *There are no data that indicate special gender distribution. Therefore, patients will be enrolled in the study gender-independently.

Exclusion Criteria:

Patients who meet any of the following criteria will be excluded from study entry:

1. Mixed cholangiocarcinoma and HCC.
2. Concurrent enrolment in another clinical study, unless it is an observational (non-interventional) study or a study without a medical intervention (specifically the PLATON registry [ClinicalTrials.gov identifier: NCT04484636] is allowed).

   Note: After the Safety Follow-up (28 days post treatment discontinuation) participation in another clinical study is allowed.
3. Major surgery (as defined by the Investigator) within 4 weeks prior to enrollment into the study; patients must have recovered from effects of any major surgery.

   Note: Local non-major surgery for palliative intent (e.g. surgery of isolated lesions, per-cutaneous biliary drainage or biliary stenting) is acceptable.
4. Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, serious active, uncontrolled, gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent.
5. History of another primary malignancy except for:

   * Malignancy treated with curative intent and with no known active disease ≥ 3 years before the first dose of IMP and of low potential risk for recurrence;
   * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease;
   * Adequately treated carcinoma in situ without evidence of disease.
6. Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to employ effective birth control from screening to 5 months after the last dose of combination therapy or for a period of at least 5 half-lives of the respective drug/IMP after the last dose of combination therapy (whichever is longer).
7. Known allergy or hypersensitivity to any of the IMPs or any of the constituents of the product.
8. Any co-existing medical condition that in the investigator's judgement will substantially increase the risk associated with the patient's participation in the study.
9. Active or History of autoimmune disease including, but not limited to, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, antiphospholipid antibody syndrome, Wegener's granulomatosis, Sjögren's syndrome, Guillain-Barré syndrome, multiple sclerosis, vasculitis, or glomerulonephritis.

Note: History of autoimmune-related hypothyroidism on a stable dose of thyroid replacement hormone, or controlled Type 1 diabetes mellitus on a stable insulin regimen may be eligible based on consultation with the sponsor. Patients with eczema, psoriasis, lichen simplex chronicus, or vitiligo with dermatologic manifestations only (e.g., patients with psoriatic arthritis are excluded) are eligible for the study provided all following conditions are met:

* Rash must cover < 10% of body surface area;
* Disease is well controlled at baseline and requires only low- potency topical corticosteroids;
* No occurrence of acute exacerbations of the underlying condition requiring psoralen plus ultraviolet A radiation, methotrexate, retinoids, biologic agents, oral calcineurin inhibitors, or high potency or oral corticosteroids within the previous 12 months.

  10. History of non-infectious pneumonitis requiring steroids, or patients with Grade ≥ 2 pneumonitis.

  11. History of active primary immunodeficiency. 12. History of allogeneic bone marrow transplantation or prior solid organ transplantation.

  13. Treatment with systemic immunosuppressive medication (including, but not limited 14. 15. to, corticosteroids, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-TNF-α agents) within 2 weeks prior to initiation of study treatment, or anticipation of need for systemic immunosuppressive medication during study treatment, with the following exceptions:
  * Patients who received acute, low-dose systemic immunosuppressant medication or a one-time pulse dose of systemic immunosuppressant medication (e.g., 48 hours of corticosteroids for a contrast allergy) are eligible for the study.
  * Patients who received mineralocorticoids (e.g., fludrocortisone), corticosteroids for chronic obstructive pulmonary disease (COPD) or asthma, or low-dose corticosteroids for orthostatic hypotension or adrenal insufficiency are eligible for the study.

    16. Administration of a live, attenuated vaccine within four weeks or for a period of at least 5 half-lives of the respective drug/IMP (whichever is longer) prior to start of enrollment, or anticipation that such a live attenuated vaccine will be required during the study or within 5 months after the last dose of atezolizumab.

    17. Significant cardiovascular disease, such as cardiac disease (New York Heart Association Class II or greater), myocardial infarction or cerebrovascular accident within 3 months prior to initiation of study treatment, unstable arrhythmias, unstable angina, and/or concurrent and clinically significant abnormalities on electrocardiogram (ECG) at Screening, including QTcF > 450 ms for males or > 460 ms for females.

    18. Clinically significant valvular defect. 19. Unable or unwilling to swallow the complete daily dose of derazantinib capsules.

    20. Clinically unstable central nervous system (CNS) metastases (to be eligible, subjects must have stable disease > 3 months, confirmed by magnetic resonance imaging (MRI) or computed tomography (CT) scan, and/or have CNS metastases well controlled by low-dose steroids, anti-epileptics, or other symptom-relieving medications).

    21. Current evidence of clinically significant corneal or retinal disorder, including but not limited to bullous/band keratopathy, keratoconjunctivitis (except for keratoconjunctivits sicca), corneal abrasion (except if related to trauma), inflammation/ulceration, confirmed by ophthalmologic examination.

    22. Significant gastrointestinal disorder(s) that could, in the opinion of the Investigator, interfere with the absorption, metabolism, or excretion of derazantinib and/or atezolizumab (e.g., Crohn's disease, ulcerative colitis, extensive gastric resection).

    23. Active tuberculosis. 24. Co-infection with hepatitis B and hepatitis C. Patients who are negative for HCV RNA will be considered non-infected for HCV.

    25. Severe bacterial, fungal, viral and/or parasitic infections on therapeutic oral or IV medication at the time of first dose of study drug administration.

    26. Treatment with strong CYP3A4 inducers within 14 days prior to initiation of study treatment, including rifampin (and its analogues) or St. John's wort.

    27. Patient who has been incarcerated or involuntarily institutionalized by court order or by the authorities § 40 Abs. 1 S. 3 Nr. 4 AMG.

    28. Patients who are unable to consent because they do not understand the nature, significance and implications of the clinical trial and therefore cannot make a rational/informed decision after receiving the study information [§ 40 Abs. 1 S. 3 Nr. 3a AMG].

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2022-04-20 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Primary Objective: Assessment of Efficacy | up to 4 years, at EOS
  Objective Response Rate (ORR) will be assessed every 8 weeks (+/- 7 days) according to RECIST 1.1 criteria

SECONDARY OUTCOMES:
Secondary Objective: Assessment of Safety | up to 4 years, at EOS
  All adverse events (including serious adverse events and adverse events of special interest) will be assessed for saftey of study treatment in accordance with CTCAE V 5.0
Secondary Objective: Assessment of Efficacy in relation to objection response rate at EOT | up to 4 years, at EOS
  Objective response rate (ORR) according to investigator-based RECIST 1.1 assessment, defined as the proportion of allocated subjects with best response of complete or partial response within study treatment.
Secondary Objective: Assessment of Efficacy in relation to progression free survival | up to 4 years, at EOS
  The proportion of patients known to be alive and without confirmed objective disease progression at 6, 8 and 10 months after first administration of study treatment, respectively and time from first administration of study treatment until the date of first objective disease progression or death.
Secondary Objective: Assessment of Efficacy in relation to overall survival | 4 years, at EOS
  Time from first administration of study treatment until death of a patient due to any cause

OTHER OUTCOMES:
Tertial Objective: Exploratory Biomarker Objective in Blood Samples | 4 years, at EOS
  Blood samples for correlative studies will be drawn at baseline, during treatment and at time of progression and samples will be used to monitor immune cell population before and during therapy.
Tertial Objective: Exploratory Biomarker Objective in Fecal Samples | 4 years, at EOS
  Fecal samples will be collected at baseline (before administration of any study medication) and on C3D1 for microbiome analysis.

CONTACTS AND LOCATIONS:
Locations (17):
- Germany (17):
  - HELIOS KLinikum Bad Saarow, Bad Saarow
  - MVZ am Oskar-Helene Heim Berlin, Berlin
  - Universitätsmedizin Berlin Charité, Berlin
  - Vivantes Klinikum Berlin Friedrichshain, Berlin
  - Johanniter Krankenhaus Bonn, Bonn
  - Uniklinikum Köln, Cologne
  - Klinikum Esslingen, Esslingen am Neckar
  - Krankenhaus Nordwest gGmbH, Frankfurt
  - Medizinische Hochschule Hannover, Hanover
  - Alexianer Krefeld GmbH, Krefeld
  - Universitätsklinikum Leipzig, Leipzig
  - Universitätsmedizin Mainz, Mainz
  - Universitätsmedizin Mannheim, Mannheim
  - LMU München Großhadern, Munich
  - Klinikum rechts der Isar, Technische Universität München, München
  - Universitätsklinikum Tübingen, Tübingen
  - Marienhospital Wesel, Wesel

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared